CLINICAL TRIAL: NCT04293432
Title: A Pharmacovigilance Study of Torsade de Pointes in the Food and Drug Administration Adverse Event Reporting System Using Data Mining Algorithms
Brief Title: A Pharmacovigilance Study of Torsade de Pointes
Status: Completed | Type: Observational
Sponsor: University of Peshawar (Other)
Responsible Party: Principal Investigator, Mohammad Ismail, Assistant Professor, Department of Pharmacy, University of Peshawar
Other Study IDs: PV-TdP
Record Dates: First submitted 2020-02-14; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Torsades de Pointe Caused by Drug
MeSH Terms: interventions — Drugs, Generic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Group/Cohort: Torsade de Pointes induced by drugs reported to the FAERS database from inception till first quarter of 2019 (1990-2019)
  Interventions: Drug: Drugs, Generic

INTERVENTIONS:
Drug: Drugs, Generic — All drugs having ≥10 TdP cases reported in the FAERS database

SUMMARY:
Many cardiac and non-cardiac drugs are associated with TdP that may constitute a significant problem because of sudden cardiac death. This study aims to present a comprehensive overview and disproportionality analysis of TdP cases reported to the Food and Drug Administration Adverse Event Reporting System (FAERS) in order to identify new signals of TdP.

DETAILED DESCRIPTION:
Drug-induced Torsade de Pointes (TdP) is a serious but an overlooked adverse drug reaction because a wide range of marketed drugs associated with TdP are commonly prescribed in routine practice. Owing to the heightened concern of a vast number of drug-TdP associations including newly approved drugs, the investigators, therefore, aims to investigate drug-TdP associations by performing disproportionality analysis in order to identify new signals of TdP utilizing the individual case reports of TdP in the FAERS database.

ELIGIBILITY:
Inclusion Criteria:

* TdP cases reported in the FAERS database till 31/03/2019
* Adverse event reported was including the MedDRA term: Torsade de Pointes

Exclusion Criteria:

* Drugs with less than 10 TdP reports

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presented with TdP treated for any disease
Sampling Method: Non-Probability Sample
Enrollment: 6670 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Identification of drugs associated with TdP | Cases reported to the FAERS database till 31/03/2019
  The search includes MedDRA (v-22) Preferred Term, "Torsade de Pointes (MedDRA code: 10044066) for the identification of all TdP case reports and drugs.
Identification of new signals of TdP | Cases reported to the FAERS database till 31/03/2019
  Signal detection using disproportionality analysis

SECONDARY OUTCOMES:
Validation of already known drug-TdP associations | Cases reported to the FAERS database till 31/03/2019
Stratification of new signals with respect to age | Cases reported to the FAERS database till 31/03/2019
Stratification of new signals with respect to gender | Cases reported to the FAERS database till 31/03/2019
Trends of TdP reports in FAERS database | Cases reported to the FAERS database till 31/03/2019
Description of the population of patients having TdP | Cases reported to the FAERS database till 31/03/2019

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacy, University of Peshawar, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ali Z, Ismail M, Rehman IU, Goh KW, Razi P, Ming LC. Association of anxiolytic drugs with Torsade de Pointes: a pharmacovigilance study of the Food and Drug Administration Adverse Event Reporting System. J Pharm Policy Pract. 2024 Sep 16;17(1):2399716. doi: 10.1080/20523211.2024.2399716. eCollection 2024. PMID 39291052